CLINICAL TRIAL: NCT04377113
Title: NK Cells, Tumor Infiltrating Lymphocytes and Cell Cytotoxicity in Renal Cell Cancer - Observational Study
Brief Title: Cellular Immunity and Renal Cell Cancer
Status: Completed | Type: Observational
Sponsor: Clinical Hospital Center Rijeka (Other)
Responsible Party: Principal Investigator, Dean Markic, Prof. of Urology, MD, PhD, FEBU, Clinical Hospital Center Rijeka
Other Study IDs: 31052020
Record Dates: First submitted 2020-05-03; First posted 2020-05-06 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2020-05

CONDITIONS: NK Cell Mediated Immunity; NK Cell Cytokine Production; Kidney Cancer
Keywords: renal cell cancer; NK cells; tumor infiltrating lymphocytes; cellular immunity
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Investigators will collect:
  1. patients with kidney cancer:
     * blood,
     * urine,
     * kidney tissue removed during operation (healthy kidney tissue, carcinomatous tissue and tissue form the border)
  2. healthy control:
     * blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- RCC patients: RCC patients (30 pts) will include patients with kidney cancer (renal cell cancer).
  Investigators will collect and analyze:
  * blood sample,
  * urine sample,
  * kidney tissue sample (healthy tissue, carcinomatous tissue and borderline tissue between them).
- Healthy patients: In this group (30 patients) will be recruiting healthy patients (volunteer).
  Investigators will collect and analyze:
  * blood sample.

SUMMARY:
Renal cell cancer (RCC) is one of the most important urogenital tumors because of it's high mortality and increasing incidence. RCC, which accounts about 3% of all malignant tumors in the adults, is the most lethal urogenital cancer. The high mortality rate stimulate investigator groups to study RCC pathogenesis including immunological part. It is interesting that immunotherapy was firstly started in patients with metastatic RCC using IL-2 and interferon gamma. The first results were promising but the exact mechanism of acting was not found. In the RCC, as in the others tumors, immune cells (T lymphocytes, NK and NKT cells) are responsible for main antitumor effect. Their effect was caused by cytotoxic activity on the tumor cells. In the investigation investigators will determine patterns of aggregation of tumor infiltrating immune cells in the blood, healthy kidney and carcinomatous tissue. But, presence of this cells not implicated that this cells are active. Their activity will be determined by proofing cytotoxicity of different subgroup of immune cells. In that way investigators will present different patterns of aggregation of tumor infiltrating immune cells and their cytotoxicity which will direct that this cells are active with antitumor effect. Correlation of collected data with classical prognostic factors in the patients with RCC as tumor staging, tumor grading (Fuhrman) and histological subtype will help to determine some immunological factors as possible new prognostic factors. For conclusion, the results of this study will allow better understanding of RCC pathogenesis, specially their immunological part and become a foundation for the future investigations.

DETAILED DESCRIPTION:
Cellular immunity will be investigated in the two group of patients: operated patients with RCC and healthy volunteers.

In the study investigators will determine patterns of aggregation of tumor infiltrating immune cells in the blood (RCC patients and volunteers), healthy kidney and carcinomatous tissue as their cytotoxicity (only RCC patients).

Investigators will determine:

1. presence of different immune cells in the blood and kidney tissue (T lymphocytes, NK cells, NKT cells, T regulatory cells),
2. presence and distribution of cytolytic molecule perforin and granulysin in immune cells (T lymphocytes, NK cells, NKT cells) in the blood, kidney tissue and urine
3. NK cytotoxicity
4. possible correlation between presence of immune cells and clinical prognostic factors

ELIGIBILITY:
Inclusion Criteria:

* RCC (renal cell cancer) patients
* operated patients
* both gender
* older than 18 years
* written informed consent

Exclusion Criteria:

* age younger of 18
* patients with metastatic disease
* patients receiving antibiotics 6 weeks before operation
* patients regularly treated with corticosteroids or immunosuppressive drugs
* transplanted patients
* patients with autoimmune diseases and/or vasculitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Two groups of the patients:
  1. Patients operated because of RCC (30 patients)
  2. Healthy volunteers (30 patients)
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2020-05-24 (Actual); Primary Completion 2021-07-26 (Actual); Study Completion 2021-07-26 (Actual)

PRIMARY OUTCOMES:
Distribution of immune cells between two groups measured in the blood samples | 7 months
  Determination of distribution of immune cells between two groups in their blood samples with their comparison.
Distribution of immune cells between different tissue samples (RCC vs. healthy tissue vs. borderline tissue) | 7 months
  Determination of distribution of immune cells between different tissue samples with their comparison
Determination of NK cytotoxicity | 7 months
  Determination of NK cytotoxicity

CONTACTS AND LOCATIONS:
Overall Officials: Dean Markić, MD, PhD, Principal Investigator — Clinical Hospital Center Rijeka
Locations (1):
- Clinical Hospital Center Rijeka, Rijeka, Croatia

IPD SHARING:
Plan to Share IPD: No
All included patients will signed informed consent. Individual participant data will not be shared with other researchers.

REFERENCES:
- [Background] Sotosek S, Sotosek Tokmadzic V, Mrakovcic-Sutic I, Tomas MI, Dominovic M, Tulic V, Sutic I, Maricic A, Sokolic J, Sustic A. Comparative study of frequency of different lymphocytes subpopulation in peripheral blood of patients with prostate cancer and benign prostatic hyperplasia. Wien Klin Wochenschr. 2011 Dec;123(23-24):718-25. doi: 10.1007/s00508-011-0096-7. Epub 2011 Nov 23. PMID 22105113
- [Background] Sotosek Tokmadzic V, Laskarin G, Mahmutefendic H, Lucin P, Mrakovcic-Sutic I, Zupan Z, Sustic A. Expression of cytolytic protein-perforin in peripheral blood lymphocytes in severe traumatic brain injured patients. Injury. 2012 May;43(5):624-31. doi: 10.1016/j.injury.2010.05.009. Epub 2010 May 26. PMID 20537642
- [Background] Mrakovcic-Sutic I, Bacic D, Golubovic S, Bacic R, Marinovic M. Cross-talk between NKT and regulatory T cells (Tregs) in modulation of immune response in patients with colorectal cancer following different pain management techniques. Coll Antropol. 2011 Sep;35 Suppl 2:57-60. PMID 22220404
- [Background] Xia Y, Zhang Q, Zhen Q, Zhao Y, Liu N, Li T, Hao Y, Zhang Y, Luo C, Wu X. Negative regulation of tumor-infiltrating NK cell in clear cell renal cell carcinoma patients through the exosomal pathway. Oncotarget. 2017 Jun 6;8(23):37783-37795. doi: 10.18632/oncotarget.16354. PMID 28384121
- [Background] Cozar JM, Canton J, Tallada M, Concha A, Cabrera T, Garrido F, Ruiz-Cabello Osuna F. Analysis of NK cells and chemokine receptors in tumor infiltrating CD4 T lymphocytes in human renal carcinomas. Cancer Immunol Immunother. 2005 Sep;54(9):858-66. doi: 10.1007/s00262-004-0646-1. Epub 2005 May 11. PMID 15887015
- [Background] Shabtai M, Ye H, Frischer Z, Martin J, Waltzer WC, Malinowski K. Increased expression of activation markers in renal cell carcinoma infiltrating lymphocytes. J Urol. 2002 Nov;168(5):2216-9. doi: 10.1016/S0022-5347(05)64358-3. PMID 12394762
- [Background] Zhang Q, Jia Q, Deng T, Song B, Li L. Heterogeneous expansion of CD4+ tumor-infiltrating T-lymphocytes in clear cell renal cell carcinomas. Biochem Biophys Res Commun. 2015 Feb 27;458(1):70-6. doi: 10.1016/j.bbrc.2015.01.069. Epub 2015 Jan 28. PMID 25637538
- [Background] Oldham KA, Parsonage G, Bhatt RI, Wallace DM, Deshmukh N, Chaudhri S, Adams DH, Lee SP. T lymphocyte recruitment into renal cell carcinoma tissue: a role for chemokine receptors CXCR3, CXCR6, CCR5, and CCR6. Eur Urol. 2012 Feb;61(2):385-94. doi: 10.1016/j.eururo.2011.10.035. Epub 2011 Nov 4. PMID 22079021
- [Background] Finke JH, Tubbs R, Connelly B, Pontes E, Montie J. Tumor-infiltrating lymphocytes in patients with renal-cell carcinoma. Ann N Y Acad Sci. 1988;532:387-94. doi: 10.1111/j.1749-6632.1988.tb36356.x. No abstract available. PMID 2972244